CLINICAL TRIAL: NCT01598064
Title: Clinical Trial of Probiotics in Preventing Complication Related to Portal Hypertension in Cirrhotic Patients
Brief Title: Probiotics for Liver Cirrhosis With Portal Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Po-Lin Chen, MD (Other)
Collaborators: Grape King Bio Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Po-Lin Chen, MD, Doctor, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GK#10
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-07

CONDITIONS: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GK#10 (Experimental): GK#10 1 pk tid for 8 weeks
  Interventions: Dietary Supplement: GK#10
- Placebo (Placebo Comparator): Placebo 1 pack tid for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: GK#10 — GK#10, 1 pack tid
  Other Names: Probiotics
  Arms: GK#10
Drug: Placebo — Placebo 1 pack tid po
  Arms: Placebo

SUMMARY:
Recent studies indicate that probiotics can stimulate intestinal immunity and tighten the junctions of epithelial cells. By these ways, probiotics can reduce bacterial translocation; hence, they can ameliorate systemic inflammatory status. Because cirrhotic patients with portal hypertension often suffer from infections from intestinal flora, the investigators speculate that probiotics will be beneficial to those patients.

DETAILED DESCRIPTION:
The investigators will recruit appropriate patients, 120 in number, randomly allocate into control and experimental arms. They will be given GK#10 or placebo for 8 weeks. Clinical parameters, such as liver function, renal function, and general conditions will be evaluated at specific time points, week 0, 5, 9, and 13 weeks. Primary outcome measurement will be survival and major complications analysis, and secondary outcome measurement will be liver function evaluation.

The investigators anticipate providing our sponsor with useful results about GK#10. The investigators will make clear the impacts from individual strains, the investigators will validate our speculation that probiotics do no harm to cirrhotic patients with portal hypertension, even be beneficial to them. If the investigators can validate the anticipation, patients can enjoy benefits from our study, and the probiotics may have the potential to sell to the patients in the world.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with history of complications related to liver cirrhosis, including hepatic encephalopathy, variceal bleeding, and spontaneous bacterial peritonitis
2. Patients with evidences of portal hypertension, such as hepatosplenomegaly, thrombocytopenia (< 100,000/ml)

Exclusion Criteria:

1. Active infection
2. Dialysis patients, myocardial infarction, life-threatening cardiac arrythmia and stroke
3. Hepatocellular carcinoma with life expectancy < 6 months
4. Portal vein thrombosis
5. in hepatic encephalopathy or liver function ALT > 3 x UNL, T-bilirubin > 4.0 mg/dL
6. GI tract bleeding in recent 1 weeks
7. Drug abuser
8. No informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Zhang Lin, Principal Investigator — Professor
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Guerrero Hernandez I, Torre Delgadillo A, Vargas Vorackova F, Uribe M. Intestinal flora, probiotics, and cirrhosis. Ann Hepatol. 2008 Apr-Jun;7(2):120-4. PMID 18626428
- [Background] De Minicis S, Brenner DA. NOX in liver fibrosis. Arch Biochem Biophys. 2007 Jun 15;462(2):266-72. doi: 10.1016/j.abb.2007.04.016. Epub 2007 May 2. PMID 17531188
- [Background] Groszmann RJ. Hyperdynamic circulation of liver disease 40 years later: pathophysiology and clinical consequences. Hepatology. 1994 Nov;20(5):1359-63. No abstract available. PMID 7927273
- [Background] Johansson ML, Molin G, Jeppsson B, Nobaek S, Ahrne S, Bengmark S. Administration of different Lactobacillus strains in fermented oatmeal soup: in vivo colonization of human intestinal mucosa and effect on the indigenous flora. Appl Environ Microbiol. 1993 Jan;59(1):15-20. doi: 10.1128/aem.59.1.15-20.1993. PMID 8439146
- [Background] Salminen S, Salminen E. Lactulose, lactic acid bacteria, intestinal microecology and mucosal protection. Scand J Gastroenterol Suppl. 1997;222:45-8. doi: 10.1080/00365521.1997.11720717. PMID 9145446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GK#10 | Placebo
Started | 25 | 24
Completed | 25 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GK#10 | Placebo | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12) | 58.9 (10.6) | 59.4 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  Taiwan | 25 | 24 | 49
Reasons of cirrhosis [Number; unit: participants]
  CIRRHOSIS UNKNOWN REASONS | 4 | 3 | 7
  CIRRHOSIS WITH REASONS | 21 | 21 | 42
Alcoholism [Number; unit: participants]
  ALCOHOLSIM | 2 | 2 | 4
  NON-ALCOHOLISM | 23 | 22 | 45
HBV [Number; unit: participants]
  HBV | 9 | 11 | 20
  NON-HBV | 16 | 13 | 29
HCV [Number; unit: participants]
  HCV | 8 | 6 | 14
  NON-HCV | 17 | 18 | 35
Ascites [Number; unit: participants]
  ASCITES | 9 | 7 | 16
  NO ASCITES | 16 | 17 | 33
Variceal bleeding [Number; unit: participants]
  VARICEAL BLEEDING | 0 | 1 | 1
  NO VARICEAL BLEEDING | 25 | 23 | 48
Hepatic encephalopathy [Number; unit: participants]
  HEPATIC ENCEPHALOPATHY | 2 | 4 | 6
  NO HEPATIC ENCEPHALOPATHY | 23 | 20 | 43
Diabetes [Number; unit: participants]
  DIABETES | 6 | 6 | 12
  NON DIABETES | 19 | 18 | 37
Hypertension [Number; unit: participants]
  HYPERTENSION | 4 | 3 | 7
  NON HYPERTENSION | 21 | 21 | 42
Cerebral vascular accident [Number; unit: participants]
  CVA | 0 | 0 | 0
  NON CVA | 25 | 24 | 49
WBC (cells/ml) [Mean (Standard Deviation); unit: cells/ml] | 5019 (2027) | 5116 (1815) | 5111 (1886)
Hb (g/dL) [Mean (Standard Deviation); unit: g/dL] | 12.8 (1.8) | 13.2 (2.1) | 13.0 (2.0)
Platelet (x1000 platelets/μl) [Mean (Standard Deviation); unit: x1000 platelets/uL] | 108.3 (58.2) | 112.3 (45.9) | 110.2 (50.5)
Cr (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.3) | 0.9 (0.2) | 0.8 (0.3)
Total bilirubin (mg/dL) [Mean (Standard Deviation); unit: mg/dL] — Bilirubin is excreted in bile and urine, and elevated levels in blood may indicate liver function impairment.
  mg/dL | 1.2 (0.6) | 1.2 (0.6) | 1.2 (0.6)
AST (U/L) [Mean (Standard Deviation); unit: U/L] | 58.4 (24.8) | 51.1 (20.9) | 54.6 (22.5)
ALT (U/L) [Mean (Standard Deviation); unit: U/L] | 48.2 (29.3) | 39.5 (21.3) | 43.6 (25.0)
Prothrombin time (seconds) [Mean (Standard Deviation); unit: seconds] — The prothrombin time are measures of the extrinsic pathway of coagulation. It is used to determine the clotting tendency of blood. The longer prothrombin time means impairment of blood coagulation.
  seconds | 12.4 (1.1) | 11.8 (1.5) | 12.3 (1.3)
hsCRP (mg/L) [Mean (Standard Deviation); unit: mg/L] | 7.1 (0.5) | 7.4 (1.3) | 7.2 (0.9)
Malondialdehyde (μM) [Mean (Standard Deviation); unit: μM] — Malondialdehyde (MDA) is one of the most frequently used indicators of lipid peroxidation, also a biomarker of oxidative stress.
  μM | 0.6 (0.2) | 0.6 (0.2) | 0.6 (0.2)
Re-admission [Number; unit: participants]
  Re-admission | 2 | 3 | 5
  No re-admission | 23 | 21 | 44
TNF-α (pg/mL) [Mean (Standard Deviation); unit: pg/mL] — Tumor necrosis factor alpha (TNF-α) is a cytokine involved in systemic inflammation and is a member of a group of cytokines that stimulate the acute phase reaction.
  pg/mL | 12.0 (3.9) | 10.8 (2.9) | 11.4 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Admission Due to Complications Related to Portal Hypertension
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | GK#10 | Placebo
Number analyzed (Participants) | 25 | 24
participants | 2 | 3
Statistical Analysis 1: Comparison: GK#10 vs Placebo; Test type: Superiority or Other; p = 0.25, Chi-squared

2. Secondary Outcome: Liver Function Evaluation
Description: Measure ALT level of patients
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- GK#10: 8 Week: GK#10 1 pack three times per day for 8 weeks, and F/U ALT level.
- Placebo: 8 Week: Placebo 1 pack three times per day for 8 weeks, and F/U ALT level.
Arm/Group | GK#10: 8 Week | Placebo: 8 Week
Number analyzed (Participants) | 16 | 19
U/L | 48.9 (30.1) | 39.2 (19.4)

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | GK#10 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No